CLINICAL TRIAL: NCT00006080
Title: Phase II Evaluation of Fenretinide NSC (374551) as a Single Agent in the Treatment of Adult Patients With Recurrent Malignant Glioma
Brief Title: Fenretinide in Treating Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NABTC-9905; CDR0000068068 (Registry Identifier: PDQ (Physician Data Query)); UCLA-0006094
Record Dates: First submitted 2000-08-03; First posted 2003-12-23 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Astrocytoma; Oligodendroglioma; Glioma | interventions — Fenretinide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: fenretinide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of fenretinide in treating patients who have recurrent malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of fenretinide as assessed by 6-month progression- free survival in patients with recurrent malignant glioma. II. Determine the rate of measurable clinical response, time to progression, and overall survival of patients treated with this drug. III. Determine the unexpected toxicity of this drug in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to disease type (glioblastoma multiforme (closed to accrual as of 05/31/2001) and gliosarcoma (closed to accrual as of 05/31/2001) vs anaplastic astrocytoma, anaplastic oligodendroglioma, and mixed malignant glioma). Patients receive oral fenretinide twice daily during weeks 1 and 4. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline and then before each course of chemotherapy. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 41-85 patients (21-45 with anaplastic astrocytoma, anaplastic oligodendroglioma, and mixed malignant glioma and 20-40 with glioblastoma multiforme (closed to accrual as of 05/31/2001) and gliosarcoma (closed to accrual as of 05/31/2001)) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed supratentorial malignant primary glioma Glioblastoma multiforme (closed to accrual as of 05/31/2001) Gliosarcoma (closed to accrual as of 05/31/2001) Anaplastic astrocytoma Anaplastic oligodendroglioma Mixed malignant gliomas Original histological diagnosis of low-grade glioma allowed if a subsequent histological diagnosis of malignant glioma is confirmed Prior treatment for no more than 2 prior relapses allowed Disease progression documented by at least 2 pre-study brain scans Recent prior tumor resection of recurrent or progressive tumor allowed if recovered from the effects of prior surgery

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: More than 8 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL (may be transfusion dependent) Hepatic: Bilirubin less than 2 times upper limit of normal (ULN) SGOT less than 2 times ULN Renal: Creatinine less than 1.5 mg/dL Creatinine clearance at least 60 mL/min Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective barrier contraception during and for at least 2 months after study Able to swallow capsules No active infection No disease or other serious concurrent medical illness that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 1 week since prior interferon At least 1 week since prior thalidomide Chemotherapy: Recovered from prior chemotherapy At least 4 weeks since prior cytotoxic therapy (2 weeks for vincristine, 3 weeks for procarbazine, or 6 weeks for nitrosoureas) Endocrine therapy: At least 1 week since prior tamoxifen Prior steroids allowed if on stable or decreasing dose for at least 5-7 days before baseline MRI If steroid dose is increased between date of baseline MRI and initiation of study drug, a new baseline MRI is required Radiotherapy: Not specified Surgery: See Disease Characteristics No concurrent surgery Other: At least 1 week since any prior noncytotoxic agents (e.g., isotretinoin) No other concurrent anticancer therapy, including other investigational drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-09-25 (Actual); Primary Completion 2004-09-14 (Actual); Study Completion 2004-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinay K. Puduvalli, MD, Study Chair — M.D. Anderson Cancer Center
Locations (11):
- United States (11):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Puduvalli VK, Yung WK, Hess KR, Kuhn JG, Groves MD, Levin VA, Zwiebel J, Chang SM, Cloughesy TF, Junck L, Wen P, Lieberman F, Conrad CA, Gilbert MR, Meyers CA, Liu V, Mehta MP, Nicholas MK, Prados M; North American Brain Tumor Consortium. Phase II study of fenretinide (NSC 374551) in adults with recurrent malignant gliomas: A North American Brain Tumor Consortium study. J Clin Oncol. 2004 Nov 1;22(21):4282-9. doi: 10.1200/JCO.2004.09.096. PMID 15514370